CLINICAL TRIAL: NCT06560658
Title: Optimizing Microdosing and Meditation
Acronym: OMM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding was obtained.
Sponsor: National University of Natural Medicine (Other)
Responsible Party: Principal Investigator, Matthew Hicks, Principial Investigator, National University of Natural Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OMM
Record Dates: First submitted 2024-08-12; First posted 2024-08-19 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Meditation; Microdosing
Keywords: psilocybin; microdosing; meditation
MeSH Terms: interventions — Psilocybin; Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Microdosing only (Experimental)
  Interventions: Drug: Psilocybin
- Microdosing plus meditation (Experimental)
  Interventions: Drug: Psilocybin; Behavioral: Meditation

INTERVENTIONS:
Drug: Psilocybin — Participants will receive four 2-hour sessions of supervised microdosing of psilocybin in a two week period.
  Other Names: psilocybin microdosing
Behavioral: Meditation — Participants will receive four 2-hour sessions of supervised microdosing of psilocybin in a two week period. In addition to meditating during their sessions, participants will also meet online five days a week for meditation instruction and practice.
  Arms: Microdosing plus meditation

SUMMARY:
The goal of this clinical trial is to test the feasibility of combining meditation with psilocybin microdosing in healthy adults. The main questions it aims to answer are:

1. Recruitment and retention feasibility
2. Acceptability, Safety and Tolerability
3. Exploratory Measures:

3.1: Explore potential changes in sleep quality and duration, heart rate variability, and other biometric outcomes captured by the Oura Ring (3rd generation).

3.2: Explore potential changes in quality of life scores 3.3: Explore potential differences in altered states of consciousness across groups 3.4: Explore qualitative data collected during sessions and at follow-up to assess satisfaction and receive feedback about the intervention.

Every participant will receive the psilocybin microdosing intervention, however, half of the participants will be randomly selected to receive the meditation intervention.

DETAILED DESCRIPTION:
Research has shown that both meditation and high doses of psilocybin can produce enhanced feelings of well-being that persist. When combined, the synergistic effects might be more than the sum of the parts when treating mental health challenges like depression. The results for microdosing, on the other hand, are mixed, and there have yet to be studies on the synergy between microdosing and meditation.

If the synergy between microdoses of psilocybin and meditation is significant, this suggests the possibility of a safe, effective, and low-cost intervention involving group-based meditation training and practice combined with a psilocybin microdosing protocol. The Oregon Psilocybin Services program provides a unique opportunity to test this possibility in the context of services now legally available to clients, allowing researchers to assess the safety and efficacy in a real-life context.

Project aims and methods This study aims to test the feasibility of the model by assessing recruitment, retention, acceptability, safety, and preliminary efficacy of the intervention. In addition to an appropriate medical screening and intake we will collect questionnaire data using the Credibility/Expectancy Questionnaire (CEQ), PROMIS-29, Five Facet of Mindfulness Questionnaire (FFMQ), Pittsburgh Sleep Quality Index (PSQI), Altered States of Consciousness (11-ASC) rating scale, and a survey and structured interview. During a one week wash-in period, the intervention period, and for one month after the intervention, Oura rings will be used to collect over 20 biometric data points including sleep quality, respiration rate, heart rate variability, and more.

Participants will consist of adults in Oregon that will be individually screened by a study investigator and then randomized into two arms. One arm will receive microdosing only consisting of one group preparation session and two microdosing sessions per week for two weeks. The other arm will receive the same microdosing protocol with the addition of morning online meditation practice Monday through Friday for both weeks, and will utilize meditation practices during their microdose sessions. The meditation sessions will include opportunities for the group to discuss their meditation experiences and a psychoeducational component to further improve outcomes. This content will provide participants with a better understanding of the ruminations that interrupt their focus while meditating and encourage greater distance from, and less distress concerning, those thoughts.

Expected outcomes The authors hypothesize that the model will be feasible if we are able to recruit at least 20 out of 24 expected participants, have an 80% retention rate of participants during the two week intervention period, participants on average rate their satisfaction of the intervention as 3.0 or higher on a 5-point scale, there are no more than ten adverse events or more than one serious adverse event, and data from exploratory measures indicate that further investigation is warranted.

Despite the U.S. Food and Drug Administration (FDA) granting Breakthrough Therapy status to psilocybin for the treatment of depression,56 it remains on the Drug Enforcement Agency's (DEA) Schedule I list of controlled substances alongside heroin and cocaine. While the DEA and the FDA have become increasingly more willing to grant waivers for research into psychedelic drugs, the proposed study does not require such a waiver to comply with the law. This is due to the unique construction of Oregon's Psilocybin Services Act (Chapter 475A of Oregon Statutes). The state law creates a program wherein licensed growers, inspected by licensed laboratories, can distribute psilocybin mushrooms to licensed service centers. It is only within the approved boundaries of these service centers and while supervised by a licensed facilitator that the mushrooms can be consumed by clients who must stay on site for a designated amount of time that depends on the dose.

According to Oregon Health Authority Administrative rule 333-333-5130, facilitators of psilocybin service are prohibited from (1) practicing any other scope of practice they may have (e.g. naturopathic medicine) while facilitating, and (2) handling, selling, or transferring psilocybin at any time. Thus, while it is technically true that growers, services centers, and clients are liable for trafficking and possession of a Schedule I substance, the federal government has adopted a policy of allowing state programs such as this in a manner similar to their policy on cannabis. Complying with Oregon law means that study investigators are not administering or providing psilocybin, but instead are studying the facilitation of the services. At the request of the Institutional Review Board (IRB) of the National University of Natural Medicine (NUNM) for a similar study, this rationale was confirmed via direct communication with the regional DEA office who agreed with this interpretation of both federal and state law. Participants are given clear information on their liability in order to provide consent.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older - Oregon Psilocybin Services Act sets the minimum eligible age of 21.
* Able to attend all study events.
* Able to read and speak fluent English.
* No more than 100 hours of lifetime meditation experience.
* No prior experience of microdosing of a psychedelic substance and no more two macrodose experiences.

Exclusion Criteria:

* A personal or family history of an immediate family member of schizophrenia, psychosis of any kind, mania, or hypomania.
* A current prescription for lithium, antipsychotic, Phase II UGT substrate such as diclofenac or probenecid, or an unwillingness to taper off these or other medications that the study clinicians determine to be a risk for interactions.
* Active suicidal ideations or history of suicide attempts. Passive ideation, such as "I wouldn't mind if I never woke up again" is permissible.
* Uncontrolled hypertension or heart disease.
* Any form of personality disorder.
* Current recreational drug use or any form of substance abuse in the previous six months.
* Pregnancy, plans to become pregnant during the study period, or breast feeding.
* Active cancer treatment.
* Any mental illness that could currently be rated as severe. This includes but is not limited to a PHQ-9 score above 20, GAD-7 score above 14, or their equivalents on comparable scales and acute trauma related symptoms.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment and Retention Feasibility | From time of approval to completion of the study, up to one year.
  Determine the recruitment rate (number of participants enrolled compared to those approached).
  Evaluate the participant retention rate throughout the study, including psilocybin sessions and follow-up assessments.
Acceptability | From time of approval to completion of the study, up to one year.
  Assess participant satisfaction with the group psilocybin-assisted therapy format through qualitative interviews and survey questions.
Safety and Tolerability | From time of approval to completion of the study, up to one year.
  Monitor the incidence and severity of adverse events associated with psilocybin administration in a group setting.

OTHER OUTCOMES:
Subjective Sleep quality and duration | Seven weeks, a one week wash-in period, two weeks during the primary intervention, and for four weeks post-intervention
  Explore potential changes in sleep quality and duration via Pittsburgh Sleep Quality Index.
Objective Sleep quality and duration | Seven weeks, a one week wash-in period, two weeks during the primary intervention, and for four weeks post-intervention
  Explore potential changes in sleep quality and duration, heart rate variability, and other biometric outcomes captured by the Oura Ring (3rd generation).
Quality of life | At four time points in a seven week period
  Explore potential changes in quality of life scores assessed by PROMIS-29 (Patient Reported Outcomes Measurement Information System), which captures seven health domains (physical functioning, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbances).
Altered states of consciousness | At each of the four microdosing sessions during the two week intervention period
  Explore potential differences in altered states of consciousness across groups using the 11-ASC (Eleven Dimensions of Altered States of Consciousness Rating Scale)
Qualitative data | Collected at all study events, up to one year.
  Qualitative data will be collected during sessions and at follow-up including comments and feedback about the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hicks, ND, MS, Principal Investigator — National University of Natural Medicine
Locations (1):
- National University of Natural Medicine, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
No data from this project is intended for any public or private repository. However, project data and relevant protocols for which no public repository exists will be made available upon request.
  We will not publish our trial protocol nor will we deposit data to public data warehouses. We will make our data and statistical code available to journal editors upon request for open access publications and/or to confirm our results.